CLINICAL TRIAL: NCT02120040
Title: Psychosocial Consequences of the Screening of Von Hippel Lindau Diseases for Patients Operated for a hémangioblastoma of Nervous Centrasl System
Acronym: PsychoVHL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-01
Record Dates: First submitted 2014-04-16; First posted 2014-04-22 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Hemangioblastoma (HB) of the Central Nervous System (CNS)
MeSH Terms: conditions — Hemangioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hemangioblastoma (HB) of the Central nervous system (CNS) (Other)
  Interventions: Other: evaluation of anxiety with psychosocial scales

INTERVENTIONS:
Other: evaluation of anxiety with psychosocial scales

SUMMARY:
Von Hippel-Lindau (VHL) disease is a severe autosomal dominant genetic disorder (with almost complete penetrance) that predisposes to many tumors including some associated with a poorer outcome. Clear cell renal cell carcinoma (CCRCC) is the leading cause of mortality.

The diagnosis of VHL disease may be challenging because tumors have an asynchronous and multi-organ development and there is often no apparent hereditary context. As it is admitted that VHL disease is underdiagnosed, some countries have decided to recall patients presenting one of the potentially VHL disease-associated tumors to screen them for VHL mutation. Screening is currently recommended in guidelines but many patients may have not been previously screened.

Hemangioblastoma (HB) of the Central nervous system (CNS) is one of the typical VHL tumors and up to 20% of patients with HB show VHL mutation. VHL diagnosis in this population enables the diagnosis of other tumor types at an early stage of development since HB is chronologically the second tumor occurring during the VHL disease history.

But it raises critical problems and questions: difficult announcement of a potentially severe disease and psychosocial dimension related to inheritance of the disease.

ELIGIBILITY:
Inclusion Criteria:

* age >=18;
* Surgery for a CNS HB in the department of Neurosurgery of la Timone university hospital since 1999 ;
* Absence of prior screening for VHL

Exclusion Criteria:

* minor,
* incorrect French language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2014-05-02 (Actual); Primary Completion 2015-10-09 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
evaluate the impact on anxiety of VHL mutation screening of patients operated for HB | two years
  The main objective of this study is to evaluate the impact on anxiety of VHL mutation screening of patients operated for HB

SECONDARY OUTCOMES:
assessment of the mood | two years
  The evaluation of the mood will be made from Beck's scale. It is about a scale allowing to make a fast self-assessment of the depression

OTHER OUTCOMES:
assesment of quality of life | two years
  The measure of the quality of life will be made by means of a generic questionnaire: the SF36. The SF36, used for the evaluation of the remote quality of life of the plan of announcement, is validated and available in French language
assesment of the psychological consequences of the screening | two years
  The psychological consequences of the screening will be estimated by means of Psychological Consequences Questionnaire . It is about a specific instrument allowing to estimate the psychosocial impact of the screening

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Metellus, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France